CLINICAL TRIAL: NCT01456702
Title: Influence of Pre-operative Risk Stratefiction and Intraoperaitve Monitoring on Perioperative Volume Therapy and Postoperative Outcome
Brief Title: Risk Stratification and Goal-directed Volume Therapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Michael Sander, Vice Chair, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: VoMo
Record Dates: First submitted 2011-09-29; First posted 2011-10-21 (Estimated); Last update posted 2013-12-31 (Estimated); Status verified 2013-12

CONDITIONS: Fluid Volume Disorder
Keywords: SVV; hemodynamic monitoring; goal-directed volume therapie

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- control arm (No Intervention): volume therapy via standard operating procedure
- intervention arm (Experimental): goal-directed volume therapy due to svv in dependence of preoperative risk stratefication
  Interventions: Procedure: risk stratification group

INTERVENTIONS:
Procedure: risk stratification group — goal-directed volume therapy due to svv measurement or volume therapy via standard operated procedures in dependence of cardiac risk factores
  Other Names: svv group
  Arms: intervention arm

SUMMARY:
It is difficulte to evaluate risk patients and to find the ideal intraoperative volume management. It seems to be that ill patients benefit of a goal directed volume management. The aim of this study is to implement the guidelines on perioperative cardiovascular evaluation and care for non-cardiac sugery and to improve perioperative a goal-directed protocoll for volume management.

DETAILED DESCRIPTION:
It is difficult in the majority of cases to estimate the correct intra-operative mass of fluid therapy for each patient und needs a high degree of clinical experience. Among circumstances and problems of surgery (kind of surgery, length of time, bleeding, loss of liquid via wound) and kind of anesthesia, are also the concomitant diseases of patients relevant for the action of all anesthetists. These concomitant diseases correct to detect and to deduce corresponding consequences calls likewise for high clinical experience. Furthermore, the pre-operative fasting is an important fact.

Considering all these influencing factors the anesthetist tends rather to apply to much volume during surgery, followed by much more problems in PACU and / or intensive care unit.

However, how much volume is correct for which patient during which kind of surgery? How could the investigators estimate the really intra vessel volume deficit? Which available parameters are helpful, which monitoring is useful? These questions confront daily every anesthetist.

Monitoring of clinical "traditional" factors such as diuresis, blood pressure und heart rate are from experience to inexactly. Actually exist in the experts no uniform opinion about the kind and amount of fluid administration, which to apply, as well as the adequate monitoring. The central venous pressure, a commonly used parameter, is falling more and more behind.

Cardiac filling pressures correlate bad with filling volume and are unsuitable parameters for fluid therapy. It seems that dynamic parameters such as stroke volume (SV) and stroke volume variation (SVV) are better markers. SV and SVV could be measured by usual invasive blood pressure via LiDCO- or FloTrac-Monitoring.

In the study the investigators would show, that it is necessary to optimize processes already in the anesthetic ambulance, to evaluate patients with theirs concomitant diseases correctly followed by an improvement of intra-operative processes.

With the help of questionnaire is to be better structured and classified the cardiac risk of patients in accordance with the actually ACC / AHA guidelines (8). Depending surgery risk, the development of intra-operative monitoring happens standardized preoperatively (NIBP vs. IBP vs. SVV via FlowTrac or LiDCO). The intra-operative fluid regime will be performing in the group of NIBP and IBP on the basis of standard operating procedures (SOP) as well as in the group of SVV on the basis of a targeted-volume protocol.

There are a lot of surgeries with an increased fluid turnover and increased risk for cardiac complication. This demonstrated study limits the kind of surgeries on orthopedic operations with different requirement of intra-operative volume.

Hypothesis The daily challenge of each anesthetic is the correctly estimate of volume status during surgery. Multiple factors such as concomitant diseases, pre-operative fluid fasting, anesthesia as well as circumstances of surgery inclusive bleeding risk have an important influence followed by difficult peri-operative management.

The aim of this study is the improvement of peri-operative fluid management due to process optimisation already in the anesthetic ambulance included cardiac risk factors of patients followed by intra-operative fluid protocol. Primary outcome parameters are administered fluid volume (including blood transfusion), and secondary measured by amount of blood loss, postoperatively frequency of PONV, delir as well as PACU and ICU stay.

The investigator believes that the investigators could reduce the intra-operative fluid volume as well as blood loss due to these process optimization followed by increase patient satisfaction. Furthermore, the investigators could possibly reduce the PACU and ICU stay.

ELIGIBILITY:
Inclusion Criteria:

* electiv orthopedic surgery with intermediate risk surgery
* signed informed consent
* >18 years

Exclusion Criteria:

* No consent for the study
* Age < 18 years
* Emergency surgery
* Pregnant women
* Jehovah's Witnesses
* Myocardial infarction in the last 4 weeks
* High-risk cardiac factors
* GOLD IV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2014-10; Primary Completion 2015-12 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
intra- and postoperative volume | surgical time + treatment time until discharched to the ward or a maximum of 10 hours

SECONDARY OUTCOMES:
treatment time in PACU, ICU, anesthetic recovery room | admission on PACU, ICU and anesthetic recovery room until a maximum of 10 hours
incidence of delirium and PONV | admission on ICU, PACU, anesthetic recovery room until discharge to the ward or a maximum of 10 hours
need of blood tranfusions | intra- and postoperative treatment time with a maximum of 10 hours postoperative
incidence of vasopressors | intra- and postoperative treatment time until a maximum of 10h postoperative

CONTACTS AND LOCATIONS:
Overall Officials: Michael Sander, MD, Principal Investigator — Dept. of Anesthesiology CCM/CVK Charité Universitätsmedizin Berlin
Locations (1):
- Department of Anesthesiology CCM/CVK Charité Universitätsmedizin Berlin, Berlin, State of Berlin, Germany